CLINICAL TRIAL: NCT03251976
Title: The Effect of a CPR Decision Aid on CPR Knowledge and Code-Status Preferences in Patients With Advanced Gynecologic Malignancies
Brief Title: CPR Decision Aid For Patients With Advanced Gynecologic Malignancies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Kerri Bevis, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: F12345678
Record Dates: First submitted 2017-08-14; First posted 2017-08-16 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Advance Care Planning
Keywords: ovarian cancer; cardiopulmonary resuscitation; end of life care; endometrial cancer; cervical cancer
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms; Uterine Cervical Neoplasms | interventions — Videotape Recording

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): video decision aid
  Interventions: Behavioral: video
- Usual care (Active Comparator)
  Interventions: Behavioral: usual care

INTERVENTIONS:
Behavioral: video — informational video
  Arms: Intervention
Behavioral: usual care — usual physician counseling on end of life care
  Arms: Usual care

SUMMARY:
The purpose of this research is to assess the effect of a cardiopulmonary resuscitation (CPR) decision aid video on CPR knowledge and end-of-life preferences in women with advanced gynecologic malignancy. We will assess the baseline CPR knowledge in our research population, gauge the improvement after viewing a decision aid video, and evaluate its effects on patient preferences regarding CPR.

ELIGIBILITY:
Inclusion Criteria:

* patients with stage III or greater cervical, ovarian, or uterine malignancies
* receiving chemotherapy at UAB gynecologic oncology infusion center

Exclusion Criteria:

* early stage gynecologic cancer
* receiving chemotherapy at a different location
* Non-English speaking
* deafness
* blindness

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-11-06 (Actual); Primary Completion 2019-05-06 (Actual); Study Completion 2019-05-06 (Actual)

PRIMARY OUTCOMES:
CPR knowledge | one month after intervention
  Patient CPR knowledge assessment score (0-4)

SECONDARY OUTCOMES:
CPR preference | baseline
  Patient CPR preference (Yes, No, Unsure)
CPR preference | one month after intervention
  Patient CPR preference (Yes, No, Unsure)
CPR knowledge | baseline
  Patient CPR knowledge assessment score (0-4)

CONTACTS AND LOCATIONS:
Overall Officials: Kerri Bevis, MD, MSPH, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No